CLINICAL TRIAL: NCT00481663
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Dose-Ranging Finding Study of Once-Daily Dosing of Sitaglipin (MK-0431) in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Brief Title: A Study of Different Doses of Sitagliptin (MK-0431) in Participants With Type 2 Diabetes Mellitus (MK-0431-014)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-014; 2007_570
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Sitagliptin 25 mg once daily (Experimental): Sitaglipin (MK-0431), 25 mg, once daily for 12 weeks, orally. Due to interim analysis of this study and another Phase IIB study, participants in this arm were switched into the 100-mg once daily arm during either the first or initiation of the second extensions study periods.
  Interventions: Drug: Sitagliptin; Drug: Rescue
- Sitagliptin 50 mg once daily (Experimental): Sitagliptin, 50 mg, once daily for 12 weeks, orally. Due to interim analysis of this study and another Phase IIB study, participants in this arm were switched into the 100-mg once daily arm during either the first or initiation of the second extensions study periods.
  Interventions: Drug: Sitagliptin; Drug: Rescue
- Sitaglipin 100 mg once daily (Experimental): Sitagliptin, 100 mg, once daily for 158 weeks, orally
  Interventions: Drug: Sitagliptin; Drug: Rescue
- Sitagliptin 50 mg twice daily (Experimental): Sitagliptin 50 mg, twice daily for 12 weeks, orally. Due to interim analysis of this study and another Phase IIB study, participants in this arm were switched into the 100-mg once daily arm during either the first or initiation of the second extensions study periods.
  Interventions: Drug: Sitagliptin; Drug: Rescue
- Placebo to Sitagliptin → Metformin (Placebo Comparator): Placebo to Sitagliptin, once daily, orally for 12 weeks. Participants randomized to the placebo treatment group during the base study were reallocated to treatment with metformin 850 mg twice daily (b.i.d., initiated with 850 mg q.d. for 4 weeks then force titrated to 850 mg b.i.d.) during either the first or initiation of the second extensions study periods.
  Interventions: Drug: Placebo to sitagliptin; Drug: Metformin; Drug: Rescue

INTERVENTIONS:
Drug: Sitagliptin
  Arms: Sitaglipin 100 mg once daily; Sitagliptin 25 mg once daily; Sitagliptin 50 mg once daily; Sitagliptin 50 mg twice daily
Drug: Placebo to sitagliptin
  Arms: Placebo to Sitagliptin → Metformin
Drug: Metformin
  Arms: Placebo to Sitagliptin → Metformin
Drug: Rescue — Patients whose FPG >240 mg/dL from Week 16 or HbA1C >8.5% from Week 25 up to (not including) Week 52 could receive rescue antihyperglycemic therapy with pioglitazone, and remain in the extension study (Extension 1). Participants were eligible for rescue with pioglitazone 30 mg (or rosiglitazone in countries where pioglitazone was not licensed) if they met the following criteria: from Week 16 and during the second extension: FPG consistently >240 mg/dL (repeated and confirmed within 3 to 7 days); from Week 52 up to (not including) Week 70: HbA1C >8%; from Week 70 up to (not including) Visit 21/Week 106: HbA1C >7.5% (Extension 2). Participants placed on rescue therapy with pioglitazone (rosiglitazone where pioglitazone is not available) in the first or second extensions were not eligible for enrollment in the third extension. Rescue therapy was not available in the third extension.

SUMMARY:
A study of different doses of MK-0431 in participants with type 2 diabetes mellitus. There have been 3 extensions to the base study (Extension 1: up to Week 52, Extension 2: up to Week 106, and Extension 3: up to Week 158). The primary hypothesis for the study is that In participants with type 2 diabetes who have inadequate glycemic control, after 12 weeks of treatment, a dose-response will be seen across once-daily doses of MK-0431 in lowering hemoglobin A1C (HbA1c).

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant women
* Fasting plasma glucose >= 130 mg/dL
* HbA1c >=6.5% and >10.0%

Exclusion Criteria:

* You have a history of type I diabetes
* You are on a weight loss program with ongoing weight loss or taking weight loss medication
* You have had surgery within 30 days
* You hvae hepatitis B or C.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2003-08-19 (Actual); Primary Completion 2004-07-21 (Actual); Study Completion 2006-05-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in HbA1C at Week 12 | Baseline and Week 12
Number of Participants Who Experienced One or More Adverse Events (AE) up to Week 14 | Up to Week 14
Number of Participants Who Experienced One or More AE up to Week 54 | Up to Week 54
Number of Participants Who Experienced One or More AE up to Week 108 | Up to Week 108
Number of Participants Who Experienced One or More AE up to Week 160 | Up to Week 160
Number of participants Who Discontinued Study Treatment Due to An AE up to Week 12 | Up to Week 12
Number of participants Who Discontinued Study Treatment Due to An AE up to Week 52 | Up to Week 52
Number of participants Who Discontinued Study Treatment Due to An AE up to Week 106 | Up to Week 106
Number of participants Who Discontinued Study Treatment Due to An AE up to Week 158 | Up to Week 158

SECONDARY OUTCOMES:
Change from Baseline in HbA1C at Week 52 | Baseline and Week 52
Change from Baseline in HbA1C at Week 106 | Baseline and Week 106
Change from Baseline in HbA1C at Week 158 | Baseline and Week 158
Change from Baseline in Fasting Plasma Glucose (FPG) at Week 12 | Baseline and Week 12
Change from Baseline in FPG at Week 52 | Baseline and Week 52
Change from Baseline in FPG at Week 106 | Baseline and Week 106
Change from Baseline in FPG at Week 158 | Baseline and Week 158
Change from Baseline in Body Weight at Week 12 | Baseline and Week 12
Change from Baseline in Body Weight at Week 52 | Baseline and Week 52
Change from Baseline in Body Weight at Week 106 | Baseline and Week 106
Change from Baseline in Body Weight at Week 158 | Baseline and Week 158
Change From Baseline in Serum Fructosamine at Week 12 | Baseline and Week 12
Change From Baseline in Daily Seven-Point Fingerstick Glucose Average at Week 12 | Baseline and Week 12
Change From Baseline in Daily Seven-Point Fingerstick Glucose Average at Week 52 | Baseline and Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Hanefeld M, Herman GA, Wu M, Mickel C, Sanchez M, Stein PP; Sitagliptin Study 014 Investigators. Once-daily sitagliptin, a dipeptidyl peptidase-4 inhibitor, for the treatment of patients with type 2 diabetes. Curr Med Res Opin. 2007 Jun;23(6):1329-39. doi: 10.1185/030079907X188152. Epub 2007 Apr 30. PMID 17559733
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html